CLINICAL TRIAL: NCT00855556
Title: Parkinson's Disease Genetics Database
Status: Terminated | Type: Observational
Why Stopped: Enrollment into this registry was not as robust as investigator envisioned. Thus, the registry was closed.
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Michael Pourfar, Principal Investigator, Northwell Health
Other Study IDs: GCRC 0171
Record Dates: First submitted 2009-02-25; First posted 2009-03-04 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA stored in TE buffer solution
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: blood draw — The blood collection is designed to obtain blood samples as a source of DNA for genotyping and to establish a plasma and serum storage repository for future assays. GCRC nurses will perform all blood draws associated with this study. The following procedures are designed to standardize sample collection:
  1. Blood will be collected with the participant in the seated position with the reclining position reserved for those with a history of fainting during blood collection.
  2. Participants will be instructed to drink plenty of water (e.g., at least 8 large glasses of water) prior to the clinic visit as this facilitates easier collection.
  3. No fasting, activity or medication restrictions are required prior to or following blood collection.
  4. Blood collection will follow completion of the questionnaires. They will be performed by a nurse or technician with documented class time and experience in phlebotomy. Technician certification will occur prior to blood collection.

SUMMARY:
The goal of the study is to develop and organize an effort to identify genes that determine an individual's risk for developing Parkinson's disease (PD).

1. To ascertain, study and establish a repository of DNA samples that will allow for the identification of known and yet-to-be-identified genetic markers associated with the development of PD.
2. To create a database with clinical, genetic (HLA, genome screen) and medical history information that will facilitate the search for PD susceptibility genes.
3. To provide a centralized DNA repository to allow for targeted studies of genetic factors contributing to the onset, heterogeneity and progression of PD.
4. To evaluate opportunities to extend the results of research to develop methods of risk prediction, prevention and therapy for PD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a diagnosis of Parkinson's Disease as determined by standard neurological criteria.
* Patients ≥18 years of age who are able to provide informed consent
* Patients ≥ 18 who are decisionally impaired for whom informed consent can be obtained by a legally authorized representative.

Exclusion Criteria:

* Patients without a diagnosis of Parkinson's Disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a diagnosis of Parkinson's Disease as determined by standard neurological criteria.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2008-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
the current protocol is for establishment of the registry only and not for particular analyses of its contents | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pourfar, MD, Principal Investigator — Northwell Health
Locations (1):
- The Feinstein Institute for Medical Research, Manhasset, New York, United States